CLINICAL TRIAL: NCT03961438
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant HIV-1 Envelope Protein ConM SOSIP.v7 gp140 Vaccine, Adjuvanted With MPLA Liposomes, in Healthy, HIV-Uninfected Adults
Brief Title: Amsterdam UMC Clinical Trial With a Native-like HIV-1 Envelope Vaccine
Acronym: ACTHIVE-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Emma Reiss, Clinical Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL69161.000.19
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: HIV-1-infection
Keywords: Neutralizing antibody responses; Antibodies; HIV-infection; Vaccine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomised in a 1:1 ratio between two treatment groups with a different dosing regimen. The randomisation will be stratified for gender.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): HIV-uninfected participants
  Interventions: Biological: ConM SOSIP.v7 gp140, adjuvanted with MPLA liposomes
- Group B (Active Comparator): HIV-uninfected participants
  Interventions: Biological: ConM SOSIP.v7 gp140, adjuvanted with MPLA liposomes

INTERVENTIONS:
Biological: ConM SOSIP.v7 gp140, adjuvanted with MPLA liposomes — Vaccine administration will be done at months 0, 2 and 6 by intramuscular injection into the deltoid muscle of the non-dominant arm. The immunogen will be used at the dosage of 100 μg and will be admixed with 500 μg MPLA formulated in liposomes.
  Other Names: Recombinant HIV-1 trimeric gp140 Env protein: ConM SOSIP.v7.
  Arms: Group A
Biological: ConM SOSIP.v7 gp140, adjuvanted with MPLA liposomes — Vaccine administration will be done at months 0, 2 and 6 by intramuscular injection into the deltoid muscle of the non-dominant arm. The immunogen will be used at the dosage of 100 μg at months 0 and 2, and 20 μg at month 6. All immunogen dosages will be admixed with 500 μg MPLA formulated in liposomes.
  Other Names: Recombinant HIV-1 trimeric gp140 Env protein: ConM SOSIP.v7.
  Arms: Group B

SUMMARY:
ACTHIVE-001 is a randomised, open-label, uncontrolled phase 1 clinical trial to determine the safety profile of the native-like HIV-1 envelope vaccine, ConM SOSIP.v7, adjuvanted with monophosphoryl lipid A (MPLA) liposomes. The study will furthermore determine the extent to which the vaccine influences the breadth of viruses neutralised by induced antibodies and the associated diversity of B and T cell responses.

The research will also investigate the effect of a within-schedule successive dose level reduction (i.e. fractional dose boosting), aimed to induce higher levels of somatic hypermutation and broadly neutralising antibodies. The primary outcome will be measurement of adverse events. Secondary and exploratory outcomes will include specific viral neutralisation activity of serum antibodies and characterisation of antigen specific blood and lymph node B and T cell responses.

DETAILED DESCRIPTION:
Human immunodeficiency virus (HIV) causes a global pandemic that affects nearly 37 million people and continues to spread at a rate of 1.8 million new infections annually. With currently only 21.7 million people on antiretroviral therapy (ART), a protective vaccine is crucial to reduce HIV spread and eliminate the pandemic. Given their protective capacity, a vaccine that induces neutralising antibodies (NAbs) against the HIV envelope protein (Env) would be a major step forwards. Nevertheless, the design of an effective NAb inducing vaccine has proven to be extremely challenging due to the instability and conformational flexibility of the trimeric Env protein. However, the development of stabilised, native-like trimeric Env proteins, termed SOSIP trimers, has revolutionised the HIV vaccine field by overcoming this obstacle.

The SOSIP prototype, BG505 SOSIP.664, was the first ever Env-based immunogen that consistently induced NAbs against neutralisation-resistant viruses in animals and BG505 trimer immunisation of non-human primates protected against BG505 virus acquisition. Yet, HIV-1 diversity is a major hurdle for generating broad protection by broadly neutralising antibodies (bNAbs). It is thought that consensus-based vaccines might be more amendable for driving neutralisation breadth, because consensus sequences contain less strain-specific antigenic determinants and are closer to individual viral strains than strains are to one another. Therefore, the native-like Env trimer ConM SOSIP.v7 gp140, used in this study, was modelled after the BG505 SOSIP.664 prototype, but based on a consensus sequence of all HIV-1 isolates in group M, responsible for the global HIV epidemic. Previous nonclinical studies in rabbits and non-human primates found the ConM SOSIP.v7 gp140 vaccine to be safe. Moreover, it induced remarkably strong autologous NAb responses and elicited modest levels of cross-neutralisation.

Bearing these promising results in mind, the investigators firstly aim to evaluate the safety and tolerability of the ConM SOSIP.v7 gp140 vaccine, adjuvanted with monophosphoryl lipid A (MPLA) liposomes, in healthy HIV-uninfected individuals. The secondary objective will be to determine whether the ConM SOSIP.v7 gp140 vaccine, adjuvanted in MPLA liposomes, is able to prime human germline (naive) B cells and drive antibody responses towards induction of NAb breadth.

The research will furthermore investigate the effect of a within-schedule successive dose level reduction (i.e. fractional dose boosting), aimed to induce higher levels of somatic hypermutation and bNAbs. It is thought that fractional dose boosting leads to competitive antigen binding in germinal centres, which results in selection and expansion of B cells with surface immunoglobulins showing the highest antigen affinity.

The immunological insights gleaned from this study will be crucial for further design refinement and clinical development. In-depth characterisation of the elicited immune response, accomplished for example by state-of-the-art 'omics techniques such as next generation sequencing (NGS) and transcriptomics, enables us to gain valuable information from just a few human trial subjects. As a part of the European AIDS Vaccine Initiative 2020 Consortium (EAVI2020), this study will aid with the objective to select and refine the best immunogens, adjuvants, prime-boost schedules and determine the impact of host factors such as gender and genetics, increasing the chance of discovery of a definitive vaccine, which most likely will be multi-component.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged between 18 and 50 years on the day of screening.
2. Willing to comply with the requirements of the protocol and available for follow-up for he planned duration of the study.
3. Willing and able to give written informed consent.
4. Willing to undergo HIV testing, risk reduction counselling and receive HIV test results, including the possibility of vaccine-induced seropositivity (VISP).
5. All female individuals engaging in sexual activity that could lead to pregnancy must commit to use an effective method of contraception for four months following Investigational Medicinal Product administration.
6. All female volunteers who are not heterosexually active at screening, must agree to utilise an effective method of contraception if they become heterosexually active.
7. All female volunteers must be willing to undergo urine pregnancy tests at designated time points.
8. All sexually active male volunteers, regardless of reproductive potential, must be willing to use an effective method of contraception (such as consistent condom use) from the day of first vaccination until at least four months after the last vaccination to avoid exposure of partners to Investigational Medicinal Product in ejaculate and to prevent conception with female partners.
9. Willing to abstain from donating blood, eggs or sperm from the day of first vaccination until at least 3 months after the end of their participation in the trial and, for those who test HIV-positive due to vaccine-induced antibodies, until the anti-HIV antibody titres become undetectable.
10. All volunteers must be registered with a general practitioner.

Exclusion Criteria:

1. Confirmed HIV-1 or HIV-2 infection (HIV Ag/Ab plus HIV RNA testing).
2. Self-reported risk for HIV exposure or STIs prior to screening.
3. If female, pregnant or planning a pregnancy during the period of enrolment until four months after the last study vaccination; or lactating.
4. Any clinically relevant medical condition that is considered in the opinion of the investigator to make the volunteer unsuitable for participation in the study (under which underlying haematological disorders, auto-immune disease, immunodeficiency, gastrointestinal, hepatic and cardiopulmonary disorders). This also includes a history of malignancy in the past five years (prior to screening) or ongoing malignancy. (Note: A history of a completely excised malignancy that is considered cured is not an exclusion).
5. Infectious disease in the six months before screening: acute and chronic hepatitis B infection (HbsAg-positive), hepatitis C infection (anti-HCV and HCV RNA positive), treatment for chronic hepatitis C infection in the past year, or active syphilis (positive chemiluminescence immunoassay (LIAISON XL), confirmed by positive RPR).
6. History of hyposplenia (anatomical or functional).
7. Bleeding disorder that was diagnosed by a physician (e.g., factor deficiency, coagulopathy or platelet disorder that requires special precautions.) (Note: A volunteer who states that he or she has easy bruising or bleeding, but does not have a formal diagnosis and has intramuscular injections and blood draws without any adverse experience, is eligible).
8. Receipt of any vaccine within 60 days of vaccination with the Investigational Medicinal Product.
9. Receipt of blood products or blood-derived products within four months of screening.
10. Participation in another clinical trial of an Investigational Medicinal Product currently, within the previous three months or expected participation during this study. Concurrent participation in an observational study, not involving medicinal products and not requiring any blood or tissue sample collection is not an exclusion criterion.
11. Prior receipt of another investigational HIV vaccine or HIV monoclonal antibody (product). (Note: receipt of placebo in a previous HIV vaccine trial will not exclude a volunteer from participation if documentation is available.)
12. Known hypersensitivity to any component of the vaccine formulation used in this trial, or severe or multiple allergies to drugs or pharmaceutical agents.
13. Positive reaction in antinuclear antibody (ANA) screen and/or subsequent anti-dsDNA and/or anti-ENA assessment; or clinically significant immunoglobulin (IgA, IgG or IgM) values.
14. Use of any medications, including over-the-counter products, which, in the opinion of the investigators, would either interfere with the study or potentially cause harm to the volunteer. Use of corticosteroids, immunosuppressants, chemotherapeutics, anti-tuberculosis or other medications considered significant by the investigator within the previous six months. The following exceptions are permitted and will not exclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis (except for steroids applied to the non-dominant upper arm); or a short course (duration of ten days or less, or a single injection) of corticosteroid for a non-chronic condition (based on investigator clinical judgment) at least two weeks prior to enrolment in this study.
15. Unable to read and speak Dutch or English to a fluency level adequate for the full comprehension of procedures required in participation and consent.
16. Active, serious infections requiring (par)enteral antibiotic, antiviral or antifungal therapy within 30 days prior to enrolment.
17. Seizure disorder: A participant who has had a seizure in the last three years prior to screening is excluded. (Not excluded: a participant with a history of seizures who has neither required medications nor had a seizure for three years).
18. Grade ≥ 1 clinically significant routine safety laboratory parameters.
19. If, in the opinion of the Principal Investigator, it is not in the best interest of the volunteer to participate in the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Adverse events | 7 days post each vaccination
  Proportion of volunteers with a ≥ grade 3 adverse event.
Adverse events | 28 days post each vaccination
  Proportion of volunteers with ≥ grade 3 and/or vaccine related adverse events.
Vaccine-related serious adverse events | 18 months
  Proportion of volunteers with vaccine-related serious adverse events.

SECONDARY OUTCOMES:
Autologous neutralising antibodies | 18 months
  Serum titres of neutralising antibodies to virus expressing ConM envelope.
Binding antibody responses | 18 months
  Proportion and magnitude of the trimer binding antibody response.
Heterologous neutralising antibodies | 18 months
  Serum titres of neutralising antibodies against additional (Tier1a/b, Tier 2) HIV-1 virus strains.
Env-specific B cell responses | 18 months
  Measurement of the magnitude and phenotype of Env-specific plasmablast, naive, germinal centre and memory B cell responses in peripheral blood mononuclear cells (PBMC) and lymph node aspirates.

OTHER OUTCOMES:
Env-specific T cell responses | 18 months
  Measurement of the magnitude and phenotype of T cell responses in peripheral blood mononuclear cells (PBMC) and lymph node aspirates.

CONTACTS AND LOCATIONS:
Overall Officials: Godelieve de Bree, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam University Medical Centers, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Results from this study will be disseminated locally and to the wider scientific community at conferences and in published open-access peer-reviewed journals, as appropriate. Any data used for publication will be fully anonymised. We plan to publish the data and hold onto the data for 20 years.
Supporting Information: Study Protocol
Time Frame: 18 months from when the study officially closes.
Access Criteria: Directly from Dr. G.J. de Bree (g.j.debree@amsterdamumc.nl)